CLINICAL TRIAL: NCT00154245
Title: A One-year, Open Label Study to Investigate the Safety and the Effect of Enteric-coated Mycophenolate Sodium (EC-MPS) in Combination With Cyclosporine Microemulsion in de Novo Kidney Transplant Recipients.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Novartis External Affairs, Novartis Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CERL080ATW01
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Kidney Transplantation
Keywords: Enteric-coated mycophenolate sodium, transplantation, de novo, cyclosporine

INTERVENTIONS:
Drug: Enteric-Coated Mycophenolate sodium (EC-MPS)

SUMMARY:
The study is a one-year prospective, open-label, safety and efficacy study. De novo renal transplant recipients will be receiving cyclosporine, 1.44g EC-MPS (720 mg b.i.d.), and corticosteroids .The study will consist of a 12-month open-label treatment period on EC-MPS.

ELIGIBILITY:
Inclusion Criteria:

Males and females aged 18-75 years. Recipients of de novo cadaveric, living unrelated or living related kidney transplants

Exclusion Criteria:

Multi-organ recipients (e.g. kidney and pancreas) or previous transplant with any organ.

Patients who are recipients of A-B-O incompatible transplants. Patients with a historical or current peak PRA of 50%. Patients with already existing antibodies against the HLA-type of the receiving transplant.

Evidence of severe liver disease (incl. abnormal liver profile i.e. AST, ALT or total bilirubin 3 times UNL).

Patients who are HIV or Hepatitis B surface antigen positive. Patients with any known hypersensitivity to mycophenolic acid, MMF, EC-MPS, other components of the formulation (e.g. lactose).

Patients with thrombocytopenia (75,000/mm3), with an absolute neutrophil count of < 1,500/mm3, and/or leukocytopenia (< 2,500/mm3), and/or hemoglobin < 6 g/dL at Screening or Baseline.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2004-01; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Graft function 6 months post transplantation

SECONDARY OUTCOMES:
Incidence of biopsy proven acute rejection, graft loss or death within 6 and 12 months post transplantation
Incidence of biopsy proven acute rejection within 6 and 12 months post transplantation
Time to first biopsy-proven acute rejection
Severity of biopsy-proven acute rejection
Graft survival and patient survival at 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis